CLINICAL TRIAL: NCT05773443
Title: A Phase IIa Multicentre Randomized Controlled Double Blind Clinical Trial to Demonstrate Clinical Efficacy on Cognitive, Neuropsychiatric and Functional Outcomes of Ambroxol in New and Early Patients With Prodromal and Mild Dementia With Lewybodies (ANeED) - Joint Effort 21: eHealth and a PPI-program in Dementia With Lewybodies (DLB)
Brief Title: ANeED Joint Effort 21: eHealth and a PPI Program in Dementia With Lewybodies (DLB)
Acronym: JointEffort21
Status: Recruiting | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Helse Fonna (Other); Helse Stavanger HF (Other Government); University Hospital, Akershus (Other); Ullevaal University Hospital (Other); Haraldsplass Deaconess Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 103362
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Dementia, Lewy Body
Keywords: dementia, lewy, wearable, sensor, digital, device, monitoring, actigraphy
MeSH Terms: conditions — Lewy Body Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ambroxol: Digital biomarkers: Oral ambroxol medication, from day 1 to study end (at 60 mg TID (day 1-7), 120 mg TID (day 8- 14), 315 mg BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550))
  Interventions: Device: Digital biomarkers
- Placebo: Digital biomarkers: Oral placebo medication, from day 1 to study end (at 60 mg TID (day 1-7), 120 mg TID (day 8- 14), 315 mg BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550)).
  Interventions: Device: Digital biomarkers
- Caregivers: Primary family caregivers to participants
  Interventions: Device: Digital biomarkers

INTERVENTIONS:
Device: Digital biomarkers — Digital application Smartwatch Sleep monitor Movement sensor EEG-sensor

SUMMARY:
The goal of the study is to develop predictive algorithms and digital biomarkers to capture disease fluctuations in (prodromal) dementia with lewybodies (DLB) patients and to improve treatment, diagnosis and prognosis of the study drug Ambroxol, used in the ANeED study. This project is an additional study to the ANeED study, registered at ClinicalTrials.gov under NCT04588285.

DETAILED DESCRIPTION:
Currently, there is no approved treatment for DLB patients, despite the increasing prevalence of DLB. As disease symptoms fluctuate between days and within-day inpatient clinic visits do not adequately capture the fluctuation in disease symptoms. Therefore there is a need for continuous registration. Additionally as DLB caregivers report a high level of caregiver distress, we extended the study to include caregivers to collect data on caregiver distress.

For these reasons, a digital application was developed to report study medicine intake and side effects. Data collection from digital sensors (smartphone, smart watch, movement sensors, an EEG/EOG/ mood sensor and a bedside sleep monitor) register DLB symptoms continuously.

To be eligible to participate in ANeED Joint Effort 21, patients and their caregivers need to be included in the ANeED study. There will be no additional inpatient clinic visits in ANeED Joint Effort 21, as measurements in between the visits are performed in-home. These measurements include cognitive tests on the smartphone and health data gathered by a smartwatch. Additionally, 2 wearable movement sensors will measure activity and sleep, a bedside sleep monitor that registers sleep disturbances, as well as an EEG-EOG-mood sensor for a duration of one week.

ELIGIBILITY:
Inclusion Criteria:

A patient is eligible when all inclusion criteria and none of the exclusion criteria are fullfilled in the ANeED study:

1. Male or female.
2. Age ≥ 50 and ≤ 85 years of age.
3. Confirmed diagnosis of Dementia with Lewy Bodies (DLB) or Mild Cognitive Impairment in DLB (DLB-MCI).
4. MMSE score>=15
5. Able and willing to provide informed consent prior to any study related assessments and procedures at screening visit 1.
6. Capable of complying with all study procedures.
7. Willing to provide blood samples for genetic analyses of APOE and GBA.
8. Willing and able to self-administer or administer by a caregiver oral ambroxol medication, from day 1 to study end (at 60 mg TID (day 1-7), 120 mg TID (day 8- 14), 315 BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550)).
9. Able to travel to the participating study site.
10. A female participant is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 consecutive months of spontaneous amenorrhea, at least 6 weeks post-surgical bilateral oophorectomy (with or without hysterectomy) or post tubal ligation. In questionable cases, menopausal status will be confirmed by demonstrating levels of follicle stimulating hormone (FSH) 25.8 - 134.8 IU/L and oestradiol < 201 pmol/l at entry.

Women of child-bearing potential must use accepted contraceptive methods (listed below), and must have a negative serum at screening visit 1 and urine pregnancy tests at subsequent visits if applicable. An additional pregnancy test will be performed, and results obtained, prior to administration of the first dose of ambroxol.

Exclusion Criteria:

1. Current treatment with anticoagulants (e.g. warfarin) that might preclude safe completion in the opinion of the Investigator.
2. Current use of investigational medicinal product or participation in another interventional clinical trial or who have done so within 30 days prior to the first dose in the current study.
3. Exposure to more than three investigational medicinal products within 12 months prior to the first dose in the current study;
4. Confirmed dysphagia that would preclude self-administration of ambroxol up to 6 tablets daily for the duration of day 1 to day 550/Month 18.
5. Significant known lower spinal malformations or other spinal abnormalities that would preclude lumbar puncture.
6. History of known sensitivity to the study medication, ambroxol or its excipients (lactose monohydrate, granulated microcrystalline cellulose, copovidone and magnesium stearate) in the opinion of the investigator that contraindicates their participation.
7. History of known rare hereditary disorders of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
8. History of illegal substance abuse, drug abuse or alcoholism in the opinion of the Investigator that would preclude participation in the study.
9. Donation of blood (one unit or 350 ml) within three months prior to receiving the first dose of the study drug.
10. Pregnant or breastfeeding; All participants of child bearing potential in the opinion of the Investigator that would preclude participation in the study and who do not agree to use double-barrier birth control or abstinence while participating in the study and for two weeks following the last dose of study drug;
11. Any clinically significant or unstable psychiatric, medical or surgical condition that in the opinion of the PI or PI-delegated clinician may put the participant at risk when participating in the study or may influence the results of the study or affect the participant's ability to take part in the study, as determined by medical history, physical examinations, electrocardiogram (ECG), or laboratory tests.

    Such conditions may include:
    1. Impaired renal function
    2. Moderate/Severe hepatic impairment
    3. A major cardiovascular event (e.g. myocardial infarction, acute coronary syndrome, decompensated congestive heart failure, pulmonary embolism, coronary revascularisation that occurred within 6 months prior to the screening visit.
    4. Major depression, delirium or psychosis not related to DLB.
    5. Metastatic cancer or terminal illness.
12. Planned major surgery or other major treatments during study period that will interfere with study-obligations.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants already included in ANeED drug trial with willingness to comply to the additional study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Digital biomarkers for diagnostic support and medication efficacy | All patient visits from start to 18 months (end of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Arvid Rongve, PhD, Principal Investigator — University of Bergen / Helse Fonna
Locations (1):
- Helse Fonna, Haugesund, Rogaland, Norway